CLINICAL TRIAL: NCT03864432
Title: An Ascending Dose, Single/Multiple Dosing, Food Effect Clinical Trial to Evaluate Pharmacokinetics, Safety and Tolerability in Healthy Subjects After Oral Administration of Gemigliptin (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL020
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 25mg SAD (Experimental)
  Interventions: Drug: Gemigliptin 25mg
- 50mg SAD (Experimental)
  Interventions: Drug: Gemigliptin 50mg
- 100mg SAD (Experimental)
  Interventions: Drug: Gemigliptin 100mg
- 50mg Multiple dosing (Experimental)
  Interventions: Drug: Gemiglptin 50mg multiple dose

INTERVENTIONS:
Drug: Gemigliptin 25mg — Gemigliptin 50mg 1/2T
  Arms: 25mg SAD
Drug: Gemigliptin 50mg — Gemigliptin 50mg 1T
  Arms: 50mg SAD
Drug: Gemigliptin 100mg — Gemigliptin 50mg 2T
  Arms: 100mg SAD
Drug: Gemiglptin 50mg multiple dose — Gemigliptin 50mg 1T * 10days
  Arms: 50mg Multiple dosing

SUMMARY:
To determine the pharmacokinetic properties, safety and tolerability of single/multiple oral administration of Gemigliptin and Food effect in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects (aged 19~45 years at the time of screening)
* Subjects weighing between 50kg (inclusive) and 90kg (exclusive), and having a body mass index (BMI) of 17.1～25.8 (inclusive of limits).
* Subjects with a fasting plasma glucose (FPG) of 70～110mg/dL (inclusive of limits) at the time of screening
* Subjects who are willing to participate in the entire study cycle and comply with the study protocol (including contraception). Subjects who can sign the written Informed Consent Form after being informed of the study procedures.

Exclusion Criteria:

* Those with a history of allergies including drug allergies (aspirin, antibiotics, etc.), or other clinically significant allergies.
* Those with diseases of the liver (including carriers of hepatitis virus), kidney, respiratory system, endocrine system, nervous system or immune system. Those with a medical history of hematology/oncology, psychiatry or cardiovascular diseases.
* Those with a medical history of gastrointestinal diseases (ulcers, Crohn's disease, etc.) or surgery (excluding simple appendectomy or hernia repair), and these situations can affect the absorption of the study drug.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
AUClast of Gemigliptin | 0h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 16h, 24h, 36h, 48h and 72h
Cmax of Gemigliptin | 0h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 16h, 24h, 36h, 48h and 72h

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Mei Liu, Principal Investigator — Shanghai Xuhui District Central Hospital
Locations (1):
- Shanghai Xuhui Central hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No